CLINICAL TRIAL: NCT00682799
Title: Serial Analysis of Chimerism in Patients With Refractory Cytopenia (RC) Transplanted With Reduced Intensity Conditioning (RIC) EWOG MDS SCT RC RIC-06
Brief Title: Serial Analysis of Chimerism in Patients With Refractory Cytopenia (RC) Transplanted With Reduced Intensity Conditioning (RIC)
Status: Completed | Type: Observational
Sponsor: Charlotte Niemeyer, MD (Other)
Responsible Party: Sponsor-Investigator, Charlotte Niemeyer, MD, Prof. Dr. Charlotte Niemeyer, MD, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Other Study IDs: EWOG MDS SCT RC RIC-06
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Refractory Cytopenia of Childhood; Reduced Intensity Conditioning (RIC); Myelodysplastic Syndrome (MDS); Hematopoietic Stem Cell Transplantation (SCT)
Keywords: RC; RIC; MDS; SCT
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hematopoietic chimerism will be investigated from PB samples. Prior to transplant 5 ml EDTA PB from patient and donor are required and will be sent to the laboratory of the Coordinating Investigator (P.B.). Post transplant PB samples (5 -10 ml EDTA blood) from day +30 (4 days), +60(4 days), +100 (7 days) and +180 (7 days) will also being sent to the laboratory of the Coordinating Investigator (P.B.) From EDTA PB cell subpopulations will be isolated and DNA will be extracted and stored for further investigations.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, non-randomized multi-center multi-national study to evaluate the chimerism measured by STR and SNP in patients with hypoplastic RC and normal karyotype transplanted with a preparative regimen of reduced intensity.

Primary objectives:

* To study hematopoietic chimerism in whole blood and different cell population (CD14, CD15, CD 56, CD3, CD19) as well as in dendritic cells and regulatory T-cells after SCT with RIC in patients with RC
* To compare the results of chimerism obtained with standard STR PCR (sensitivity 1%) with those obtained with SNP PCR (sensitivity 0.1- 0.01%)

Secondary objectives:

* To evaluate the relationship between mixed chimerism and hematological engraftment, OS and EFS
* To study the impact of mixed chimerism in plasmacytoid dendritic and regulatory T-cells on the incidence of acute and chronic GVHD

DETAILED DESCRIPTION:
Research Question 3.1.1 Chimerism and post transplant outcome During the past 3 decades, SCT has become a well established treatment procedure for many malignant and hematopoietic disorders in children and adults.1-8 After transplantation, it has been of central interest whether the newly developed hematopoietic system is of recipient or donor origin. The investigations of the genotypic origin of post transplant hematopoiesis are called chimerism analysis. Originally, it was believed that complete donor hematopoiesis is essential to maintain engraftment after allogeneic SCT in humans.9 In the last decades, however, it became evident that donor and recipient hematopoiesis could coexist after allo-SCT in the recipient. This state of coexistence of hematopoietic cells is called mixed chimerism which might end in an "autologous recovery". In patients with refractory cytopenia SCT after myeloablative conditioning regimen allowed prompt and sustained engraftment in virtually all patients. In this disease relapse has become a very rare event. Consequently, transplant related mortality and long term squeals have become major obstacles yet to be overcome to improve the children's well being and the prognosis of the disease. In SCT with RIC, the reduction of early and late toxicity may be counterbalanced by delayed engraftment, graft rejection, mixed chimerism and GVHD.

Graft rejection It is well known that less myeloablative conditioning regimens predispose for a higher rate of mixed chimerism. Consequently, graft rejection or non engraftment is a major cause of treatment failure.

Sensitization to minor histocompatibility antigens by prior transfusions of blood products can increase this risk. The rapid development of complete chimerism in NK-cells and T-cells seems to play an important role to achieve sustained engraftment specifically in patients transplanted with a dose reduced preparative regimen. Therefore, it is important to elucidate the development of post transplant chimerism in different cell subpopulations. This will allow following and documenting proper engraftment, and will detect early hints of ongoing graft rejection.

Graft versus host disease The occurrence of GVHD is influenced by many well known factors. Although the use of nonmyeloablative SCT can reduce the severity of GVHD, GVHD remains a major complication. In our pilot study using the reduced intensity preparative regimen in RC, the probability for developing GVHD grade IIIV was 0.48. It is accepted that in comparison to myeloablative SCT, in reduced intensity preparative regimens higher proportions of host immune hematopoietic cells may persist. While donor-derived alloreactive lymphocytes are being infused, these autologous cells might possibly serve as host antigen presentation for continuous stimulation of donor T-cells. Consequently, it was speculated by the group Shapira and Slavin10 that GVHD may be similarly amplified by reduced conditioning followed by intentional administration of host cells. This hypothesis was tested in a preclinical animal model. Increased incidence of GVHD, higher mortality and increased levels of chimerism were observed in recipients reconstituted with additional host cells, particularly with non-irradiated spleen cells. Graft-versus-Leukaemia (GVL) effect was not impaired by post transplant cell administration. These results suggested that GVHD may be amplified by recipient cell infusion using either irradiated or viable stimulatory host cells. This could possibly explain the higher than anticipated incidence of GVHD and consequently the rapid displacement of host cells with conversion to 100% donor type cells in reduced intensity SCT. The present study will therefore investigate whether autologous antigen presenting cells (Auto-APC) do survive the conditioning regimen and favour to occurrence of GVHD.

ELIGIBILITY:
Inclusion Criteria:

RC patients enrolled in this study are to meet the following Inclusion Criteria:

* RC Patients with hypocellular BM normal karyotype included in the EWOG-MDS 2006 protocol who receive SCT from a MFD or a compatible (8/8) or one allelic mismatch UD
* Written informed consent by the caretakers and whenever possible the patient's assent.
* Age less than 18 years The caretakers will have given their written informed consent to participate in the study. Consent will be documented by the caretaker's dated signature which will be also signed and dated by the investigator in the participating center. If the patient is able to understand the meaning and consequences of the study and its procedures his/her written informed assent is also needed. Written informed consent has to be obtained prior to enrollment into the study.

Exclusion Criteria:

Patients who do not fulfill the Inclusion Criteria may not be included into study. Specific Exclusion Criteria are:

•Transplanted with a preparative regimen other than thiotepa, fludarabine

Max Age: 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will only be allowed to enter the trial if they or their caretakers provide written informed consent about their participation (following full explanation of the trial) and if the physician has verified that the patient meets all of the Inclusion Criteria and none of the Exclusion Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2007-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To study hematopoietic chimerism in whole blood and different cell population (CD14, CD15, CD 56, CD3, CD19) as well as in dendritic cells and regulatory T-cells after SCT with RIC in patients with RC | 5 years
To compare the results of chimerism obtained with standard STR PCR (sensitivity 1%) with those obtained with SNP PCR (sensitivity 0.1- 0.01%) | 5 years

SECONDARY OUTCOMES:
To evaluate the relationship between mixed chimerism and hematological engraftment, OS and EFS | 5 years
To study the impact of mixed chimerism in plasmacytoid dendritic and regulatory T-cells on the incidence of acute and chronic GVHD | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bader, M.D., Principal Investigator — University Children´s Hospital Frankfurt am Main
Locations (1):
- University Children´s Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Homepage of the EWOG-MDS-Study Group — http://www.ewog-mds.org